CLINICAL TRIAL: NCT00833157
Title: Effect of Glucosamine or Ibuprofen Combined With Physical Training in Patients With Knee-Osteoarthritis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Bispebjerg Hospital (Other)
Collaborators: Lund University (Other); The Danish Rheumatism Association (Other); Ministry of the Interior and Health, Denmark (Other Government)
Responsible Party: Susanne G. Petersen, doctor, Institute of Sports Medicine Copenhagen, Bispebjerg Hospital, Denmark
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: HIM-037; KF-01-18904
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2009-01-30 (Estimated); Status verified 2009-01

CONDITIONS: Osteoarthritis of the Knee
Keywords: Knee Osteoarthritis; exercise; strength training; Glucosamine; Dietary supplement; Ibuprofen; NSAID
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity | interventions — Glucosamine; Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Glucosamine (Experimental)
  Interventions: Drug: glucosamine sulphate
- Ibuprofen (Experimental)
  Interventions: Drug: ibuprofen
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: glucosamine sulphate — Subjects are administered glucosamine-sulphate tablets of 500 mg * 3 daily, while they are performing a strength-training program with both legs (*3 weekly) for 12 weeks.
  Other Names: glucosamine from Ferrosan
  Arms: Glucosamine
Drug: ibuprofen — Subjects are administered 600 mg * 2 daily, while they are performing a strength-training program with both legs (*3 weekly) for 12 weeks
  Other Names: "Ibumetin" from Nycomed (vnr:38 83 71)
  Arms: Ibuprofen
Drug: placebo — Subjects are administered placebo tablets, while they are performing a strength-training program (*3 weekly) with both legs for 12 weeks
  Arms: Placebo

SUMMARY:
The investigators will investigate the effect of glucosamine or ibuprofen combined with 12 weeks of muscle strength-training in patients with knee-osteoarthritis.

The investigators would like to elucidate whether treatment with glucosamine or NSAID interact with the effects of exercise in osteoarthritis patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 to 70 years
* Bilateral tibiofemoral osteoarthritis of the knee on x-ray
* American College of Rheumatology (ACR) clinical classification criteria

Exclusion Criteria:

* Severe health problems such as cardiovascular disease, active cancer, diabetes, kidney or liver diseases
* Excess alcohol use (> 21 alcoholic drinks per week)
* Severe overweight (BMI > 35)
* History of injury or operation in the knee, planned knee-joint replacement, other rheumatologic diseases, previous gastric ulcer, allergy to the contents of ibuprofen or glucosamine, regular strength training prior to the inclusion

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2005-02; Primary Completion 2007-07 (Actual); Study Completion 2009-03 (Estimated)

PRIMARY OUTCOMES:
muscle strength and hypertrophy | We measure before and after 12-weeks strength training.
cartilage biomarkers | We measure before and after 12 weeks strength training

SECONDARY OUTCOMES:
muscle regeneration and function | We measure before and after 12-weeks strength training.

CONTACTS AND LOCATIONS:
Overall Officials: Susanne G Petersen, MD, Principal Investigator — Bispebjerg Hospital, Institute of Sports Medicine Copenhagen

REFERENCES:
- [Derived] Petersen SG, Beyer N, Hansen M, Holm L, Aagaard P, Mackey AL, Kjaer M. Nonsteroidal anti-inflammatory drug or glucosamine reduced pain and improved muscle strength with resistance training in a randomized controlled trial of knee osteoarthritis patients. Arch Phys Med Rehabil. 2011 Aug;92(8):1185-93. doi: 10.1016/j.apmr.2011.03.009. PMID 21807137
- [Derived] Petersen SG, Saxne T, Heinegard D, Hansen M, Holm L, Koskinen S, Stordal C, Christensen H, Aagaard P, Kjaer M. Glucosamine but not ibuprofen alters cartilage turnover in osteoarthritis patients in response to physical training. Osteoarthritis Cartilage. 2010 Jan;18(1):34-40. doi: 10.1016/j.joca.2009.07.004. Epub 2009 Jul 15. PMID 19679221